CLINICAL TRIAL: NCT02970786
Title: Phase I Trial: 68Ga-NODAGA-E(c[RGDyK])2 Positron Emission Tomography for Imaging Angiogenesis in Primary and Metastatic Tumor Lesions in Humans
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Malene Martini Clausen, Principal Investigator, MD, PhD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AK-2015-1
Record Dates: First submitted 2016-11-15; First posted 2016-11-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Neuroendocrine Carcinoma; Breast Cancer; Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 68Ga-NODAGA-E(c[RGDyK])2 PET (Experimental): One injection of 68Ga-NODAGA-E(c[RGDyK])2 PET (app. 200 MBq) followed by 3 PET/CT scans 10 minutes, 1 hour and 2 hours post injection
  Interventions: Drug: Injection of 68Ga-NODAGA-E(c[RGDyK])2

INTERVENTIONS:
Drug: Injection of 68Ga-NODAGA-E(c[RGDyK])2 — Following one injection of 68Ga-NODAGA-E(c[RGDyK])2 the patients will be PET scanned at 10 minutes, 1 hour and 2 hours post injection

SUMMARY:
The primary objective of the trial is to test the new radio tracer 68Ga-NODAGA-E[c(RGDyK)]2 for PET imaging of angiogenesis. The tracer has the potential of identifying tumors with a high level of angiogenesis, which is one of the cancer hallmarks. Furthermore, the tracer can potentially be used in early response assessment to anti-angiogenic treatment.

This is a first-in-man study to test the radio tracer in cancer patients. Safety, biodistribution and dosimetry will be evaluated by repeated PET imaging (10 minutes, 1 hour and 2 hours post injection).

DETAILED DESCRIPTION:
The primary objective of the trial is to test the new radio tracer 68Ga-NODAGA-E[c(RGDyK)]2 for PET imaging of angiogenesis. The tracer has the potential of identifying tumors with a high level of angiogenesis, which is one of the cancer hallmarks. Furthermore, the tracer can potentially be used in early response assessment to anti-angiogenic treatment.

This is a first-in-man study to test the radio tracer in cancer patients. Safety, biodistribution and dosimetry will be evaluated by repeated PET imaging (10 minutes, 1 hour and 2 hours post injection).

The primary end points are safety, biodistribution and dosimetry of 68Ga-NODAGA-E[c(RGDyK)]2. In addition, the quantitative uptake of 68Ga-NODAGA-E[c(RGDyK)]2 will be compared to the expression of integrin αvβ3 measured directly in tumor tissue obtained by surgery or biopsies. The study will be monitored and evaluated in accordance with the principles of Good Clinical Practice (GCP).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with neuroendocrine cancer, breast cancer or ovarian cancer
* Capable of understanding and giving full informed consent

Exclusion Criteria:

* Pregnancy
* Lactation
* Obesity (weight above 140 kg)
* Claustrophobia

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Biodistribution | 2 hours
  Change in biodistribution estimated by PET
Dosimetry | 2 hours
  Dosimetry will be calculated with the use of OLINDA/EXM software (mSv) based on repeated PET imaging with the radiotracer 68Ga-NODAGA-E(c[RGDyK])2.
Safety of 68Ga-NODAGA-E(c[RGDyK])2 PET as measured by the number of participants with adverse events and significant changes in vital signs, electrocardiogram, and laboratory data. | 48 hours

SECONDARY OUTCOMES:
Quantitative uptake of the radiotracer 68Ga-NODAGA-E(c[RGDyK])2 in tumor tissue | 2 hours
  The patients will be PET scanned 10 minutes, 1 hour and 2 hours post injection of the radiotracer 68Ga-NODAGA-E(c[RGDyK])2. These timepoints will be used for assessment of tumor uptake by the use of maximum and mean standardized uptake value (SUV).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Physiology, Nuclear Medicine and PET, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No